CLINICAL TRIAL: NCT07088965
Title: Musculoskeletal Disorders of Postgraduate Dentistry Students and Specialist Dentists
Status: Recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Serdar Kilinc, assistant professor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-SK-12
Record Dates: First submitted 2025-07-18; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Musculoskeletal Diseases; Work-related Injury
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postgraduate Dentistry Students and Specialist Dentists: Postgraduate Dentistry Students and Specialist Dentists will be recruited.
  Interventions: Other: 16 / 5.000 survey application

INTERVENTIONS:
Other: 16 / 5.000 survey application — Participants will be administered a self-administered questionnaire containing basic demographic information, questions on job profile and lifestyle practices, as well as the Standardized Nordic Questionnaire (SNA).

SUMMARY:
This study aimed to assess the prevalence of MSDs and the level of ergonomics knowledge among dentists who are specializing in different branches or have completed specialist training.

DETAILED DESCRIPTION:
Musculoskeletal disorders (MSDs) are defined by the World Health Organization (WHO) as disorders of the muscles, tendons, peripheral nerves, or vascular systems that are not directly caused by an acute or sudden event. Painful disorders of the musculoskeletal system resulting from movements in work activities are referred to as work-related musculoskeletal disorders (WMSDs) and are often associated with a lack of recovery time and strenuous repetition. Implementing the strict rules and precautions outlined in ergonomic guidelines is essential to prevent the onset of MSDs.

MSDs are one of the most common occupational disorders among dentists. The dental profession can be physically and mentally demanding due to the numerous therapeutic procedures and the need for concentration during treatment sessions.

Therefore, this study aimed to assess the prevalence of MSDs and the level of ergonomics knowledge among dentists who are specializing in different branches or have completed specialist training. The null hypothesis was established as there is no difference in the prevalence of SSB and ergonomics knowledge level among dentists specializing in different branches.

ELIGIBILITY:
Inclusion Criteria

* Being between 25 and 60 years of age
* Having a stable professional career

Exclusion Criteria

* Having physical conditions such as rheumatoid arthritis or fibromyalgia
* Being retired
* Being an undergraduate student
* Having a history of any major accident, trauma, or medical condition causing permanent musculoskeletal disability

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Postgraduate Dentistry Students and Specialist Dentists will be recruited.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Standardized Nordic Questionnaire | Baseline
  The Standardized Nordic Musculoskeletal Questionnaire is a self-administered tool that investigates musculoskeletal symptoms (pain, discomfort, numbness) in nine anatomical regions over three time periods: the past 12 months, the past 7 days, and the day of the survey. A body chart illustrating these regions - neck, shoulders, upper back, lower back, elbows, wrists/hands, hips/thighs, knees, and ankles/feet - is used, and responses are recorded as yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)